CLINICAL TRIAL: NCT04589819
Title: Fracture Recovery for Returning to Duty (Teriparatide STRONG)
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Eisenhower Army Medical Center (U.S. Federal Agency); Moncrief Army Health Clinic (Unknown)
Responsible Party: Principal Investigator, J. Benjamin Jackson III, MD, MBA, Clinical Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-08190; NCT04533984 (obsolete NCT alias)
Record Dates: First submitted 2020-09-24; First posted 2020-10-19 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Stress Fracture of Tibia or Fibula
MeSH Terms: interventions — Teriparatide

STUDY DESIGN:
Intervention Model Description: There will be a 1:1 randomization into either the placebo arm or the 20mg teriparatide treatment arm. Soldiers will then receive training on how to self-administer study medication in a supervised setting. Both arms will receive 500mg of supplemental calcium to take orally, daily. They will then be released for the four week convalescent leave.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double-blinded study. All investigators will have access to the subjects results/outcomes, but will not know which randomization group the subject is in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Teriparatide (Active Comparator): Study participants will be randomized into either the study medication arm or a placebo arm. The study medication Forteo (teriparatide [rDNA origin] injection) (El-Lilly, Indiana, USA), will be administered via an blinded injection pen in the abdominal wall or thigh as described in the product guide. Subjects in the teriparatide arm will receive a 20mg dose of the medication daily via self-injection.
  Interventions: Drug: Teriparatide
- Placebo (Placebo Comparator): The placebo will be administered in a replica, blinded, injection pen in the same fashion. The study participant will self-administer the medication after being given a teaching session on medication administration by the study nurse.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Teriparatide — Teriparatide, an injectable synthetic parathyroid hormone, will be tested to evaluate its efficacy for decreasing the convalescence after a diaphyseal tibial stress fracture, a specific bone stress injury.
  Other Names: Forteo
  Arms: Teriparatide
Drug: Placebos — Placebo will be a sugar solution of the manufacturer's design.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The project goals are to improve combat readiness of U.S. Soldiers and sustain the availability of the military to deploy by, 1) decreasing the number of days not physically ready for duty after diagnosis of a diaphyseal tibial stress fracture, 2) decreasing the need for a physical profile or medical discharge board after bone stress injury, and 3) decreasing the recurrence rates of bone stress injuries.

DETAILED DESCRIPTION:
The study will examine the utility of a novel, non-operative, anabolic bone agent in the treatment of diaphyseal tibial stress fractures (DTSF). Teriparatide has been well studied in basic science and clinical studies to conclude its positive effects on building bone mass and preventing fractures in post-menopausal women. This allowed the medication to gain it an FDA indication for treatment in these groups. The investigators seek to explore additional uses for this anabolic agent in an at risk study population that has an imbalance of bone stress and bone formation resulting in a bone stress injury (BSI).

The only prior study to examine the effect of teriparatide on fracture healing demonstrated an absolute difference in the time to heal a fracture in the treatment groups, but was under powered to detect a difference. Given these positive results members of the research team have used these findings to administer teriparatide at the 20mg dose to young adult NCAA collegiate athletes who have DTSFs and other BSIs. The promising preliminary clinical observations have led the investigators to hypothesize that teriparatide will have a positive effect on bone healing and return to duty among service members with DTSFs.

A powered, prospective, controlled randomized study design will be utilized. Study subjects are to be recruited from the basic training corps at Fort Jackson via convenience sample. Soldiers who experience pain in the mid-shaft of the tibia during basic training will be evaluated and diagnosed according to the standard of care. Based on direct discussions with physical therapists stationed at Fort Jackson this diagnosis is often made by using a combination of bone scan and plain radiographs. After diagnosis, soldiers with a DTSF present to the physical therapy department for treatment and guidance for their progression of activities.

ELIGIBILITY:
Inclusion Criteria:

* Soldiers actively enlisted in the U.S. Army attached to basic training unit at Fort Jackson
* Soldiers diagnosed with a tibial diaphyseal BSI requiring convalescent leave
* Skeletally mature
* Willing to self-administer study medication
* Desire to continue their military commitment

Exclusion Criteria:

* History of any form of cancer
* Currently pregnant
* Paget's disease of bone
* Unexplained elevations of alkaline phosphatase (elevations in alkaline phosphatase may signal undiagnosed Paget's disease of bone)
* Pediatric and young adult patients with open epiphyses
* Prior external beam or implant radiation therapy involving the skeleton
* Recent (within the last 6 months) urolithiasis (kidney stones)
* Elevated serum calcium, alkaline phosphatase or uric acid
* Orthostatic hypotension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Time from diagnosis to full return to activity | 3 years
  Time to full return to activity will be measured in days from diagnosis of a bone stress injury to obtaining a passing Army Combat Fitness Test (ACFT) score.
Evaluation of long-term effects of the administration of teriparatide | 3 years
  The investigators will evaluate the long-term effects of the administration of teriparatide by following the study enrollees for a 1-year period after the completion of the study drug. The team will determine the incidence of drug related side effects. This data will be based on study nurse records during drug administration and from their data contained in the participants' Electronic Medical Records.
Evaluation of long-term effects of the administration of teriparatide on injury recurrence | 3 years
  The investigators will evaluate the long-term effects of the administration of teriparatide by following the study enrollees for a 1-year period after the completion of the study drug. The team will determine the incidence of injury recurrence as defined by lost duty time.
Evaluation of long-term effects of the administration of teriparatide on recurrent bone stress injury | 3 years
  The investigators will evaluate the long-term effects of the administration of teriparatide by following the study enrollees for a 1-year period after the completion of the study drug. The team will determine the incidence of additional or recurrent bone stress injury. This will be defined as a diagnosed bone stress injury by a physician, advanced practice provider or PCM (primary care manager) utilizing radiographic studies including: plain radiograph, MRI, and/or bone scan.

CONTACTS AND LOCATIONS:
Overall Officials: James B Jackson, MD, Principal Investigator — University of South Carolina School of Medicine
Locations (1):
- Fort Jackson, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The case records from this study will be available for review by members of the Institutional Review Board (IRB) at Eisenhower Army Medical Center, Fort Gordon, GA, by representatives of the Food and Drug Administration (FDA) and other governmental agencies as part of their normal duties. This study is being conducted in conjunction with faculty in the Department of Orthopedics, School of Medicine, and the Department of Exercise Science, Arnold School of Public Health at the University of South Carolina, who will also have access to the testing outcomes. All records will be kept in a confidential form. Otherwise, only the Physical Therapists and Physicians conducting this study will have access to the records from this study.